CLINICAL TRIAL: NCT06066619
Title: Can Cranberry Juice Enhance the Cognition and Motor Accuracy During Multitasking and Alleviate Some Negative Mental and Physiological Consequences of Intense Multitasking in Healthy Adults?
Brief Title: Can Cranberry Juice Enhance the Cognition Accuracy and Alleviate Negative Mental Consequences During Multitasking?
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: A coding error of testing beverages was discovered by study team
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202300950
Record Dates: First submitted 2023-09-05; First posted 2023-10-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Stress Response; Multitasking Behavior; Mental Stress; Physiological Stress; Cognitive Symptom; Motor Activity
MeSH Terms: conditions — Fractures, Stress; Multitasking Behavior; Stress, Psychological; Neurobehavioral Manifestations; Motor Activity

STUDY DESIGN:
Intervention Model Description: A total of 126 healthy participants will be recruited. Inclusion criteria includes body weight ≥110 pounds, age 30-55, BMI 18.9-29.9 kg/m^2, and education level high school and above. A stratified block randomization will be applied to separate participants into three different beverage groups. Three-digit codes will be assigned to different beverages. This coding process should be conducted by an individual who is not involved in the study. Maintain blinding by using the coded treatment labels during the study can help to eliminate potential biases in the assessment of outcomes.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cranberry Juice A (Experimental): Cranberry juice A
  Interventions: Dietary Supplement: Cranberry Juice A
- Cranberry juice B (Experimental): Cranberry juice B
  Interventions: Dietary Supplement: Cranberry Juice B
- Placebo juice (Placebo Comparator): Placebo juice that matches the appearance, taste, and calories of the treatment juices.
  Interventions: Dietary Supplement: Placebo Juice

INTERVENTIONS:
Dietary Supplement: Cranberry Juice A — Cranberry juices will be provided by Ocean Spray Company.
  Arms: Cranberry Juice A
Dietary Supplement: Cranberry Juice B — Cranberry juices will be provided from Ocean Spray Company.
  Arms: Cranberry juice B
Dietary Supplement: Placebo Juice — Placebo juice will be provided from Ocean Spray Company to match the appearance, taste, and calories of the cranberry juice.
  Arms: Placebo juice

SUMMARY:
This clinical trial aims to investigate the effects of a 70-day consumption of cranberry juice on cognitive and motor accuracy, mental and physiological stress, and stress response in healthy men and women between the ages of 30 and 55 who engage in multitasking. The trial will utilize a randomized, double-blinded, placebo-controlled design. It is worth noting that studies have shown that over half of middle-aged Americans experience stress, which can lead to cognitive decline and depression. Previous clinical trials have indicated that consuming polyphenol-rich foods can have positive effects on cognitive function in humans. However, no study to date has examined the long-term effects of cranberry juice consumption on cognitive performance, mental stress, and stress response specifically in individuals engaged in multitasking. Based on this gap in knowledge, the investigators hypothesize the following: (1) chronic consumption of cranberry juice will improve cognitive and motor accuracy, as well as mental and psychological stress responses in young adults subjected to intense multitasking. (2) cranberry juice consumption will alleviate the negative consequences of frequent intense multitasking, such as fatigue, mood fluctuations, cognitive impairment, and memory issues. Additionally, it is expected to have a positive impact on stress biomarkers and neurotransmitter levels. By conducting this clinical trial, the investigators aim to shed light on the potential benefits of cranberry juice consumption in improving cognitive performance, mitigating mental stress, and positively influencing stress responses in individuals who engage in intense multitasking.

DETAILED DESCRIPTION:
Recruitment Process (Screening Process):

Potential participants who have expressed interest in participating in the study will need to complete the recruitment process (or screening process). The recruitment process contains four questionnaires: Beck's Anxiety Inventory, Beck's Depression Inventory, Columbia-Suicide Severity Rating Scale, and Screening Questionnaire. The investigators will meticulously review these questionnaires to assess the eligibility of potential participants. Potential participants who meet the criteria for participation will be invited to a Consent visit (V1) to sign the consent form formally. Conversely, if potential participants do not meet the study's qualifications, the investigators will promptly communicate the results and securely dispose of the questionnaires containing their personal information.

There will be a total of three visits (V1, V2, and V3) in this study.

* V1: Consent visit
* V2: Baseline visit
* V3: Final visit

Participants who have completed the recruitment process and are qualified for the study will need to visit the lab in person and complete the consent process (V1). During V1, participants will have enough time to complete the consent. If the participants have any questions or concerns, the investigators will provide them with the necessary information and clarification. Also, the investigators will schedule the V2 and V3 with the participants. Upon signing the consent form, participants will enter the run-in phase of the study.

Run-in phase (Day -20 - Day 0):

• Participants will start to follow the dietary restriction.

Baseline visit (V2) & final visit (V3) (Day 0 - Day 70)

1. Participants will visit the lab on the last day of the run-in period.
2. Participants need to fast (10 h) before the blood collection.
3. Participants need to provide fecal samples.
4. Participants will complete a 24-hour food record by The Automated Self-Administered 24-Hour Dietary Assessment Tool and a dietary questionnaire on a computer.
5. Participants' body height and weight will be measured.
6. A phlebotomist will collect participants' fasting blood (20 mL).
7. Participants will be served a standardized breakfast with a cup of water (V2) or assigned juice (V3).
8. Tasks participants are going to complete:

   1. Multitasking tasks (Participants will count backward, first by 3 (Series 1), then by 7 (Series 2), and finally by 17 (Series 3) from a randomly chosen number within the 800 to 999 range. At the same time, participants will encounter rapidly diminishing dots on a computer screen and use a mouse to click on these dots as they appear. There will be a total of three series of tasks, each lasting 4 minutes, with 90-second breaks provided between each series. The entire session will span 15 minutes in total), State-trait anxiety inventory state, VAMS, heart rate, galvanic skin response, and saliva sample collection.
   2. NIH toolbox tests for cognition memory, attention, and learning ability.
   3. Assessment of emotional well-being, mental resilience, and sleep quality, and monitor participants' frustration levels, anxiety traits, mood fluctuations, stress levels, and depressive and suicidal tendencies.

V2 only: after all the tests, participants are free to leave the lab with two weeks' supply of assigned beverages (8 oz/per bottle and one bottle per day). Participants will return to the lab every other week to pick up cranberry or placebo juice. Participants will also return the empty bottle and report to study coordinators if there are any side effects or other issues. A compliance calendar will be provided to participants to remind their dietary restrictions and schedule. A token of appreciation will be given to participants every four weeks to reward compliance.

V3 only: after all the tests, participants are free to leave the lab, and their study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥110 pounds;
* Age 30-55;
* BMI 18.9-29.9 kg/m^2;
* Education level high school and above

Exclusion Criteria:

1. Heavy caffeine user (>300 mg caffeine/day or more than 2 cups of coffee/day);
2. Alcohol consumption (>3 alcohol/week);
3. Smoking (≥10 years);
4. Taking cannabis products;
5. Uncontrolled hypertension;
6. Clinically diagnosed illnesses, such as diabetes, cardiovascular disease, neurological disorders, and mental diseases;
7. Taking medications (antibiotics, etc.) that may influence study outcomes;
8. Taking vitamin/mineral supplements and are not willing to stop for the duration of the study;
9. Have specific dietary restriction (prevent from consuming the standardized breakfast or dinner sandwiches);
10. Inability to perform multitasking;
11. Inability to do blood collection on arm;
12. Inability to being video recorded while performing multitasking;
13. Inability to comply with dietary restrictions for the entire duration of the study;
14. Beck's depression inventory score of ≥21 during screening;
15. Beck's anxiety inventory score ≥21 during screening;
16. Severe suicidal tendencies (≥2);
17. Having seasonal depression;
18. Pregnancy;
19. Breast-feeding;
20. Female participants will do four pregnancy tests and their menstruation cycle need to be recorded. Female participants who do not wish to do pregnancy tests or record their menstruation cycle will be excluded.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | In baseline visit, for 15 minutes during multitasking; in final visit, for 15 minutes during multitasking. Through study completion, an average of 2 years.
  Heart rate (bpm) will be measured during multitasking.
Galvanic Skin Response | In baseline visit, for 15 minutes during multitasking; in final visit, for 15 minutes during multitasking. Through study completion, an average of 2 years.
  Galvanic skin response (micro-Siemens) will be measured during multitasking.
Salivary alpha-amylase activity | Through study completion, an average of 2 years.
  Salivary alpha-amylase activity will be assessed using ELISA kit.
Salivary cortisol level | Through study completion, an average of 2 years.
  Salivary cortisol level will be measured by an enzyme immunoassay with the Cortisol Elisa Assay Kit.
1. Assessment of Anxiety | During the recruitment process (screening process), potential participants are required to take 3-5 minutes to complete the BAI. Through study completion, an average of 2 years.
  Beck's Anxiety Inventory (BAI): presence and intensity of anxiety-related thoughts. During the recruitment process (screening process), potential participants who are having Beck's anxiety inventory score ≥21 will be excluded from this study.
  A higher score means a higher level of anxiety.
  Minimum Value: 0 Maximum Value: 63
2. Assessment of Anxiety | During the baseline and final visits, participants are required to take 3-5 minutes to complete the STAI state and STAI trait. Through study completion, an average of 2 years.
  State-Trait Anxiety Inventory (STAI):
  1. STAI anxiety state (STAI state): the current feeling of anxiety;
  2. STAI anxiety trait (STAI trait): the personality trait of anxiety.
  A higher score means a higher level of anxiety.
  Minimum Value: 20 Maximum Value: 80
1. Assessment of Mood | During the baseline and final visits, participants are required to take 3-5 minutes to complete the MFS after NIH toolbox tests. Through study completion, an average of 2 years.
  Mental fatigue scale (MFS): mental fatigue.
  A higher score means a higher level of mental fatigue.
  Minimum Value: 0 Maximum Value: 42
2. Assessment of Mood | During the baseline and final visits, participants are required to take 3-5 minutes to complete the VAMS after NIH toolbox tests. Through study completion, an average of 2 years.
  Visual analog mood scales (VAMS): the current mood.
  A higher score means a higher level of alert. A higher score means a higher level of inattentive. A higher score means a higher level of strong. A higher score means a higher level of weak. A higher score means a higher level of well-coordinated. A higher score means a higher level of disorganized. A higher score means a higher level of lethargic. A higher score means a higher level of energetic. A higher score means a higher level of incompetent. A higher score means a higher level of competent. A higher score means a higher level of happy. A higher score means a higher level of sad. A higher score means a higher level of interested. A higher score means a higher level of bored. A higher score means a higher level of mentally slow. A higher score means a higher level of quick-witted.
  Minimum Value: 0 Maximum Value: 100
Assessment of Depression | Participants are required to take 3-5 minutes to complete the BDI during recruitment process, baseline, and final visits. Through study completion, an average of 2 years.
  Beck's depression inventory (BDI): the feeling of depression. During the recruitment process (screening process), potential participants who are having Beck's depression inventory score ≥21 will be excluded from this study.
  A higher score means a higher level of depression.
  Minimum Value: 0 Maximum Value: 63
Assessment of Stress | During the baseline and final visits, participants are required to take 3-5 minutes to complete the PSS after NIH toolbox tests. Through study completion, an average of 2 years.
  Perceived stress scale (PSS): the feeling of stress.
  A higher score means a higher level of stress.
  Minimum Value: 0 Maximum Value: 40
Sleep Assessment | During the baseline and final visits, participants are required to take 3-5 minutes to complete the LSE after NIH toolbox tests. Through study completion, an average of 2 years.
  Leeds sleep evaluation (LSE): sleep assessment.
  Participants will place marks on a group of 10-cm lines representing they have experienced in variety of symptoms of sleep. Lines extend between extremes like "more difficult than usual" and "easier than usual". Responses are measured using a 100-mm scale and are then averaged to provide a score for each domain. Theses can then be used to evaluate the efficacy and sleep-related side effects of juices.
Suicide Severity Assessment | During the recruitment process, baseline, and final visits, participants are required to take 2 minutes to complete the CSSRS. Through study completion, an average of 2 years.
  Columbia-Suicide Severity Rating Scale (CSSRS): suicide severity rating. During the recruitment process (screening process), potential participants who are having CSSRS (answer YES to actually having thoughts about killing yourself and thinking about you might do this) will be excluded from this study. Also, appropriate actions will be taken to ensure participants safety and well-being. For example, immediately contact a specified consultant and refer the participants who with high level of suicidality to the Crisis Hot Line. Suicidal assessments will also be assessed in V2 and V3 to ensure the participants do not have any suicidal tendencies. In sum, the assessment of suicidal should be completed immediately following the completion of the instruments.
Picture Vocabulary Test | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the Picture Vocabulary Test. Through study completion, an average of 2 years.
  NIH Toolbox Picture Vocabulary Test: to assess participants' ability to understand and identify the meaning of words by matching them to corresponding images.
Flanker Inhibitory Control and Attention Test | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the Flanker Inhibitory Control and Attention Test. Through study completion, an average of 2 years.
  NIH Toolbox Flanker Inhibitory Control and Attention Test: to assess participants' cognitive control and attentional processes, specifically their ability to inhibit irrelevant information and focus on the relevant stimuli.
List Sorting Working Memory Test | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the List Sorting Working Memory Test. Through study completion, an average of 2 years.
  NIH Toolbox List Sorting Working Memory Test: to assess participants' working memory abilities.
Dimensional Changes Card Sort Test | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the Dimensional Changes Card Sort Test. Through study completion, an average of 2 years.
  NIH Toolbox Dimensional Changes Card Sort Test: to assess the cognitive flexibility of participants.
Pattern Comparison Processing Speed Test | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the Pattern Comparison Processing Speed Test. Through study completion, an average of 2 years.
  NIH Toolbox Pattern Comparison Processing Speed Test: to assess the cognition processing speed of participants.
Picture Sequence Memory Test | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the Picture Sequence Memory Test. Through study completion, an average of 2 years.
  NIH Toolbox Picture Sequence Memory Test: to assess participants' episodic memory.
Auditory Verbal Learning Test | During the baseline and final visits, participants are required to take about 40-50 minutes to complete the Auditory Verbal Learning Test. Through study completion, an average of 2 years.
  Auditory Verbal Learning Test: to assess participants' attention, memory, and learning ability in the auditory-verbal domain.
Fecal Content of Acetic acid, Propionic acid, and Butyric acid | Participants are required to provide their fecal samples on the baseline and final visit. Through study completion, an average of 2 years. Through study completion, an average of 2 years.
  Fecal content of acetic acid, propionic acid, and butyric acid will be determined using gas chromatography with a flame ionization detector.
Brain-derived neurotrophic factor (BDNF) Levels in Plasma | A certified nurse will perform a blood draw for participants during both the baseline and final visits, using two tubes, resulting in a total of 20 mL. Through study completion, an average of 2 years.
  BDNF levels in plasma will be measured using ELISA kit.
Neurotransmitters Analysis | A certified nurse will perform a blood draw for participants during both the baseline and final visits, using two tubes, resulting in a total of 20 mL. Through study completion, an average of 2 years.
  Monoamine oxidase (MAO) activity in plasma will be determined using the Amplex Red MAO Assay Kit.
1. Neurotransmitters Analysis | A certified nurse will perform a blood draw for participants during both the baseline and final visits, using two tubes, resulting in a total of 20 mL. Through study completion, an average of 2 years.
  Plasma levels of tryptophan metabolites (3-indole propionic acid, Indole-3-aldehyde , Serotonin, and Melatonin) will be quantified using the targeted metabolomic method.
2. Neurotransmitters Analysis | A certified nurse will perform a blood draw for participants during both the baseline and final visits, using two tubes, resulting in a total of 20 mL. Through study completion, an average of 2 years.
  Plasma levels of catecholamines (Dopamine, Epinephrine, and Norepinephrine) will be quantified using the targeted metabolomic method.
3. Neurotransmitters Analysis | A certified nurse will perform a blood draw for participants during both the baseline and final visits, using two tubes, resulting in a total of 20 mL. Through study completion, an average of 2 years.
  Plasma levels of histamine will be quantified using the targeted metabolomic method.
4. Neurotransmitters Analysis | A certified nurse will perform a blood draw for participants during both the baseline and final visits, using two tubes, resulting in a total of 20 mL. Through study completion, an average of 2 years.
  Plasma levels of Gamma-Aminobutyric acid (GABA) will be quantified using the targeted metabolomic method.
24-Hour Food Record | During the baseline and final visits, participants are required to take about 10-15 minutes to complete the 24-Hour Food Record. Through study completion, an average of 2 years.
  24-hour dietary record will be completed by participants using an Automated Self-Administered Dietary Assessment Tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Food/Environment Toxicology Lab, Gainesville, Florida, United States